CLINICAL TRIAL: NCT05419648
Title: Role of Monocytes Sub-populations in Thrombosis Associated With Myeloproliferative Neoplasms (MonSThr)
Acronym: MonSThr
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/29
Record Dates: First submitted 2022-06-02; First posted 2022-06-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myeloproliferative Neoplasm
Keywords: Myeloproliferative Neoplasms; Thrombosis; Monocytes sub-populations; Flow cytometry
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PV and ET patients: For the main objective, the cohort will be composed of PV and ET patients, some with a history of thrombosis and some without any history of thrombosis. A comparison will also be performed between patients with different MPN (PV or ET) and different driver mutation (JAK2V617F, JAK2 exon 12, CALR, MPL or absence of such mutations)
  Interventions: Biological: 1 additional tube of blood

INTERVENTIONS:
Biological: 1 additional tube of blood — For all the patients included, a specific blood sampling will be performed in addition to the classical evaluations that are performed in routine practice

SUMMARY:
Myeloproliferative neoplasms (MPN) are hematological malignancies associated with a major risk of thrombosis. Monocytes are hematopoietic cells with a central role in thrombosis. An activation of monocytes has been demonstrated in MPN patients. However, their study in MPN and their thrombotic complications has never been performed. In this study, we aim to evaluate the association between monocytes sub-populations and thrombotic risk in MPN patients.

DETAILED DESCRIPTION:
Myeloproliferative Neoplasms (MPN) are hematological malignancies characterized by an increased risk of thrombosis, in particular in Polycythemia Vera (PV) and Essential Thrombocythemia (ET). Predicting the risk of thrombosis in PV and ET patients helps at determining their care (use of antiaggregant and cytoreductive therapies), but relies only on limited clinical and biological criteria (age over 60 years, history of thrombosis, presence of the JAK2V617F mutation, presence of cardiovascular risk factors). Monocytes sub-populations could represent a new biomarker of thrombotic risk in PV and ET patients. Indeed, it has been shown that monocytes are activated and exhibit pro-thrombotic properties in MPN patients, especially those with a history of thrombosis. Some studies have suggested the CD16+ monocytes (intermediate and non-classical monocytes) are associated with an increased risk of arterial thrombosis. Because these monocytes are observed in inflammatory contexts, and because MPN are associated with a chronic inflammation, MPN could be associated with an increase of the proportion or the absolute count of CD16+ monocytes that could be involved in thrombotic complications observed in PV and ET patients.

In this project, an association between the proportion of CD16+ monocytes and thrombosis in PV and ET patients will be searched. Monocytes sub-populations will be studied in PV and ET patients at diagnosis as described by Selimoglu-Buet et al.1 The proportion of CD16+ (intermediate + non-classical) monocytes will be compared between patients presenting with a history of thrombosis and those without any history of thrombosis. The association between the absolute count and the proportion of CD16+, intermediate and non-classical monocytes and the occurrence of thrombosis before diagnosis, the MPN phenotype, the driver mutation, the allelic burden, the clinico-biological presentation and the existence of an inflammatory state will also be evaluated. Due to the low frequency and the high latency of thrombosis reoccurrence, patients' samples only at diagnosis (or during the year after diagnosis) will be analyzed and an association with a history of thrombosis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (age ≥ 18 years)
* Inclusion at diagnosis or during the year following the diagnosis of PV or ET (2016 WHO criteria except bone marrow biopsy that is optional in the presence of a marker of clonality)
* Subject registered with a social security scheme
* Written informed consent obtained

Exclusion Criteria:

* Patients with cytoreductive treatment (hydroxyurea, anagrelide, interferon, ruxolitinib) at the time of blood sampling
* Chronic inflammatory disease (cancer, vasculitis, rheumatism, hepato-gastro-intestinal diseases).
* Long term anti-inflammatory treatments:

  * Corticoids
  * Nonsteroidal anti-inflammatory drugs
  * Aspirin (> 325 mg per day)
  * Cyclo-oxygenase II inhibitors
* Persons under judicial safeguards, trustee or curatorship
* Person unable to give her consent
* Non-cooperative person
* Exclusion period after another clinical study or participation to another clinical study in the 30 days before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Polycythemia Vera (PV) or Essential Thrombocythemia (ET), the 2 Myeloproliferative Neoplasms (MPN) most associated with a risk of thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
History of thrombosis | At inclusion, up to 1 year after diagnosis
  Patients wil be classified as having a history of thrombosis if they had a deep vein thrombosis, pulmonary embolism, splanchnic thombosis or any other significant thrombosis. Tinnitus, vertigo, headaches, erythromelalgia as well as superficial vein thrombosis will not be considered as thrombotic events

SECONDARY OUTCOMES:
Proportion of CD16+ monocytes in PV and ET patients | At inclusion, up to 1 year after diagnosis
  The proportion of CD16+ monocytes will be assessed in PV and ET patients, and compared between patients with a history of thrombosis and those without any history of thrombosis
Proportion of monocytes sub-populations | At inclusion, up to 1 year after diagnosis
  The different sub-populations will be defined according to the expression profile of CD14 and CD16, defining classical monocytes (CD14++CD16-), non-classical monocytes (CD14loCD16++) and intermediate monocytes (CD14+CD16+). The proportion of these sub-populations will be assessed in PV and ET patients, and compared between patients with a history of thrombosis and those without any history of thrombosis
Count of monocytes sub-populations | At inclusion, up to 1 year after diagnosis
  The count (G/L) of the different monocytes sub-populations, ie CD16+ monocytes, classical monocytes (CD14++CD16-), non-classical monocytes (CD14loCD16++) and intermediate monocytes (CD14+CD16+) will be assessed in PV and ET patients, and compared between patients with a history of thrombosis and those without any history of thrombosis
Type of MPN | At inclusion, up to 1 year after diagnosis
  The type of MPN will be determined according to the WHO criteria as PV or ET. Patients will be classified as PV if they have an increased hemoglobin level (>16.5g/dL for men, >16g/dL for women), hematocrit (>49% for men, >48% for women), or red cell mass (>125% of theoretical value), together with a mutation in the JAK2 gene (JAK2V617F or exon 12), and a subnormal EPO level. If performed, bone marrow biopsy should be in favor of an MPN.
  Patients will be classified as ET if they present a thrombocytosis > 450 G/L, with a detectable mutation in JAK2, CALR or MPL. If performed, bone marrow biopsy should be in favor of an MPN.
Driver mutation of MPN | At inclusion, up to 1 year after diagnosis
  At diagnosis, a driver mutation is searched in MPN patients. We will classify patients in different groups depending on whether they carry the JAK2V617F mutation, a mutation in JAK2 exon 12, a mutation in CALR exon 9, a mutation in MPL exon 10 or any of these mutations (triple negative category). We will thus distinguish 5 groups of patients: "JAK2V617F", "JAK2 exon 12", "CALR exon 9", "MPL exon 10", "triple negative". The proportion of monocytes sub-populations will be compared between these different groups of patients
Hemoglobin level | At inclusion, up to 1 year after diagnosis
  A correlation between the hemoglobin level (g/dL) and monocytes sub-populations proportion will be searched
Platelets level | At inclusion, up to 1 year after diagnosis
  A correlation between the platelets level (G/L) and monocytes sub-populations proportion will be searched
Leukocytes level | At inclusion, up to 1 year after diagnosis
  A correlation between the leukocytes level (G/L) and monocytes sub-populations proportion will be searched
Thrombosis risk factors | At inclusion, up to 1 year after diagnosis
  A correlation between the proportion or count of monocytes sub-populations and thrombosis risk factors will be searched. These include age>60 years, history of thrombosis, tobaccoe use (actual or stopped for les than 3 years), hyperLDLcholesterol level (LDL-Cholesterol > 3,36 mmol/L), hypoHDLcholesterol level (HDL < 1,03 mmol/L in men or < 1,29 mmol/L in women), diabetes (glycemia > 6,93 mmol/L), high blood pressure (> 140/90 mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MANSIER, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux, Hématologie clinique et thérapie cellulaire, Bordeaux
  - CHU de Bordeaux, Laboratoire Hématologie, Bordeaux
  - CHU de Bordeaux, Médecine interne et immunologie clinique, Bordeaux
  - CHU de Bordeaux, Médecine Interne et maladies infectieuses, Bordeaux
  - Institut Begonié, Hématologie clinique, Bordeaux

IPD SHARING:
Plan to Share IPD: No